CLINICAL TRIAL: NCT04948216
Title: Management and Healthcare Utilization of Patients With COPD and Asthma During the COVID-19 Epidemic in Beijing
Brief Title: Management and Healthcare Utilization of Patients With Chronic Airway Disease During the COVID-19 Epidemic
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Sun Yongchang, Head of Respiratory and Critical Care Medicine, Peking University Third Hospital
Other Study IDs: LM2020133
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
During the COVID-19 epidemic, the medical treatment, disease status, and medication status of patients with chronic airway disease have not been studied. The purpose of this study is to investigate the management and healthcare utilization of patients with chronic airway disease and the influencing factors during the COVID-19 epidemic.

DETAILED DESCRIPTION:
During the COVID-19 epidemic, the medical treatment, disease status, and medication status of patients with chronic airway disease have not been studied. The purpose of this study is to investigate the management and healthcare utilization of patients with chronic airway disease and the relevant factors during the COVID-19 epidemic. Using cross-sectional research methods, telephone interviews and questionnaire surveys were used to investigate the management and healthcare utilization of patients with chronic airway disease （COPD and asthma）during the COVID-19 epidemic.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients and asthma patients in the Chronic Airway Disease Database in Peking University Third Hospital.

Exclusion Criteria:

* Refusal to participate in this study; cognitive dysfunction.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the database were involved.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Respiratory symptoms | through study completion, an average of 2 week.
  COPD Assessment Test (CAT)
Frequency of exacerbation during the COVID-19 epidemic | through study completion, an average of 2 week.
  Frequency of exacerbation during the COVID-19 epidemic

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Sun, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China